CLINICAL TRIAL: NCT02588690
Title: Beauty from Within Community Screening Project
Acronym: BFW
Status: Active, not recruiting | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Noel Bairey Merz, Director, Cedars-Sinai Medical Center
Other Study IDs: Pro00041183
Record Dates: First submitted 2015-10-19; First posted 2015-10-28 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Heart Health Screening and Prevention

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Women participating in screening: Community screening project targets women of color and/or low income women over 21 years of age in economically and ethnically diverse greater Los Angeles community. Women will be risk stratified based on ASCVD risk calculation and if labeled high risk will be referred to physician services. In 1 year, women will have their ASCVD re-risk stratify to see if seeing a physician/ health care provider reduced overall ASCVD risk scores.
  Interventions: Procedure: Fingerstick cholesterol test; Other: Atherosclerosis Cardiovascular Disease Risk assessment; Procedure: Blood pressure measurement

INTERVENTIONS:
Procedure: Fingerstick cholesterol test — A finger stick draws approximately four drops of blood. The total cholesterol (TC), High Density Lipoprotein Cholesterol (HDL-C), Triglycerides, Low Density Cholesterol (LDL-C), and Glucose tests are done.
Other: Atherosclerosis Cardiovascular Disease Risk assessment — This Risk Estimator enables estimation of 10-year and lifetime risks for atherosclerotic cardiovascular disease (ASCVD), defined as coronary death or nonfatal myocardial infarction, or fatal or nonfatal stroke, based on the Pooled Cohort Equations and lifetime risk prediction tools. The Risk Estimator is intended for use in those without ASCVD with a LDL-cholesterol <190 mg/dL.
  The information required to estimate ASCVD risk includes age, sex, race, total cholesterol, HDL cholesterol, systolic blood pressure, blood pressure lowering medication use, diabetes status, and smoking status.
  Other Names: ASCVD Risk Score
Procedure: Blood pressure measurement — Blood pressure measurement

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of death world-wide in women. Despite current medical advances, heart disease is rising in relatively young women. Women access primary care differently than men, most utilizing their Obstetrics-gynecology clinic for primary care services. The recent implementation of the Affordable Care Act (ACA) aims to provide increased access to primary care services, however, women are still not appropriately risk stratified for CVD disease risk. Many women still are not aware that they are at risk for CVD. This is particularly true for the 15-44 year old female age group. Lack of proper risk stratification may be related to women not being properly identified or appropriately referred to preventive cardiovascular services for treatment of traditional risk factors such as diabetes, obesity, hypertension, and dyslipidemia. These traditional risk markers serve as examples of chronic diseases, which are not always recognized in the early stages and therefore not optimally managed. Furthermore, if women are not feeling ill, they are less likely to access their current primary care resources for preventive strategies. Investigators propose to risk stratify women in places where they usually congregate. In addition to convenience, current risk stratification is improved with the recent implementation of the ASCVD risk calculator. Investigators hypothesize that if women were properly risk stratified and referred to appropriate preventive cardiovascular risk clinics, more preventive strategies could be implemented, therefore reducing the amount of unnecessary premature disease in women. To achieve this ambitious goal, investigators propose a three step, demonstration project.

The specific aims of this proposal is to:

1. Provide women with CVD risk stratification in places where they locally convene on a daily basis.
2. To evaluate the efficacy of a lay professional to adequately assess CVD risk.
3. To evaluate if assessment of CVD risk reduces the amount of future CVD (unsure if this can be measured in this project).

The specific aims:

1. Demonstrate feasibility and acceptability of strategies utilizing ASCVD risk assessment.
2. Improve ASCVD risk scores one year follow-up.
3. Increase heart disease awareness through marketing materials in women in Los Angeles.
4. Develop preliminary feasibility and efficacy data for a large clinical outcome trial.

DETAILED DESCRIPTION:
ACTIVITIES PLANNED FOR OCTOBER 2015 THROUGH DECEMBER 2015

1. October 2015: The Barbra Streisand Women's Heart Center (BSWHC) research team will work closely with the Preventive Cardiovascular Nurses Association (PCNA), Los Angeles (LA) Chapter as well as the community partners will develop a detailed, comprehensive screening, education, referral and ASCVD tool kit. The tool kit will include a basic demographic screening questionnaire, smart-phone ASCVD risk calculator software, cholestech finger stick supplies, blood pressure equipment, Heart Truth program materials, and Red dress pins. Educational materials developed by all partners for each community highlighting Heart Truth branding will be included. A list and specific contacts for proximate California Affordable Care Act (ACA) Community Medical Homes will be included.
2. October 2015: 2 women heart disease patient volunteers from Central and/or East Los Angeles will travel to the Mayo Clinic through the WomenHeart Program for public speaking and peer group leadership training.
3. November 2015: The 88th Street Temple Church in central Los Angeles will help develop a detailed screening tool kit with training, educational materials and collaboration with Cedars-Sinai Medical Center (CSMC) staff to perform 100 ASCVD risk assessments after church services.
4. DECEMBER 2015: The Hadassah Zionist Women's Group, Los Angeles Chapter will host a mall walking event targeting Orthodox Jewish women for screening. They will help develop a detailed screening tool kit with training, educational materials and collaboration by CSMC staff to perform 100 ASCVD risk assessments.

ACTIVITIES PLANNED FOR JANUARY 2016 THROUGH MAY 2016

1. February 2016: The CSMC Heart Truth, Wear Red Day Event: Our 2015 Heart Truth/Wear Red Day event had over 600 attendees and screened 200 women CSMC employees. If funded, the 2016 program will be open to the public.
2. February 2016: Beauty Shop Screenings. 3 local nursing organization chapters (Hispanic Nurses Society Los Angeles Chapter, Black Nurses Society LA Chapter, and Philippine Nurses Association of Southern California) will individually host a screening day in a community hair salon for at least 100 women at each site. This project is modeled after the National Heart, Lung, and Blood Institute (NHLBI)-sponsored Cedars-Sinai (CS) Barber-1 project which demonstrated blood pressure reduction in African American men using their barber as health educator. Each organization will receive a screening tool kit with training, educational materials and collaboration with CSMC staff.
3. May 2016: CSMC Telemundo Community Outreach Program. Nearly 1,500 Latino women were screened last year at the CSMC Telemundo event. The investigators will utilize the screening tool kit with intensive training, educational materials and close collaboration with CSMC staff. The theme of the 2016 event will be The Heart Truth: for women by women.
4. May 2016: Mother's Day Dinner and Health Fair at Jordan Downs Housing Development. CSMC Coach for Kids will host an annual Mother's Day Dinner for approximately 200 women at the Jordan Downs (public) Housing Development in Central Los Angeles. The community is low-income with approximately 50% African American and 50% Latino ethnicity. A health lecture (presented in both English and Spanish) and a health fair will utilize the detailed screening tool kit with Heart Truth materials.

ELIGIBILITY:
Inclusion Criteria:

* women over the age of 21

Exclusion Criteria:

* Children under the age of 21 years
* Pregnant women

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community screening project targets women of color and/or low income women in economically and ethnically diverse greater Los Angeles community
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2015-11; Primary Completion 2030-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
ASCVD Risk Score | One year
  Comparing ASCVD Risk Score calculated during initial visit and a score calculated in one year.

CONTACTS AND LOCATIONS:
Overall Officials: C.Noel Bairey Merz, MD, FACC, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Women's Heart Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes